CLINICAL TRIAL: NCT01089582
Title: Quality Of Life Assessment In AD Patients Receiving Aricept Tablets (Donepezil Hydrochloride)
Brief Title: Quality Of Life Assessment In Alzheimer's Disease (AD) Patients Receiving Aricept Tablets
Acronym: QUEST
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A2501054
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Results first posted 2010-08-03 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Alzheimer Disease
Keywords: non-interventional; mild to moderate Alzheimer's; ARICEPT.
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AD patients
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This study assessed the Hr QoL (Health related Quality of life) of subjects with mild to moderate AD, who received ARICEPT under usual clinical practice.

DETAILED DESCRIPTION:
This non-interventional study enrolled patients with mild to moderate dementia of the Alzheimer's type, who have been prescribed treatment with ARICEPT under usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's Disease

Exclusion Criteria:

* There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild to moderate dementia of the Alzheimer's type
Sampling Method: Non-Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- Greece (29):
  - University Hospital of Alexandroupolis Dimokritio, Alexandroupoli, Thrace
  - General Hospital of Arta, Arta
  - NIMITS (Geriatric Department), Athens
  - NIMITS Geriatric Department, Athens
  - General Hospital of Athens Laikon Dementia Department, Athens
  - Naval Hospital, Dementia Department, Athens
  - General State Hospital "G. Genimatas", Neurology Department, Athens
  - ATTIKON University General Hospital (Dementia Department), Athens
  - Psychiatric Hospital of Attica Dromokaiteio, Psychiatric Department, Athens
  - 1st IKA Hospital Neurology Clinic, Athens
  - Sismanogleio Psychiatric Clinic, Athens
  - HYGEIA Diagnostic & Therapeutic Center of Athens Internal Medicine Department, Athens
  - 251 General air force hospital, Athens
  - Psychiatric Hospital, Psychogeriatric Clinic, Chaïdári
  - Venizeleio General Hospital, Crete
  - Hospital of Chania, Crete
  - Hospital of Giannitsa, Giannitsá
  - University General Hospital, Ioannina
  - General Hospital of Ioannina, Ioannina
  - Center of Psychiatric Health of Katerini, Katerini
  - General Hospital Neurological Clinic, Kavala
  - Ag. Andreas, Pátrai
  - A.H.E.P.A University General Hospital of Thessaloniki, Thessaloniki
  - B´ IKA Panagia Hospital, Dementia Departments, Thessaloniki
  - Papageorgiou hospital, Thessaloniki
  - Psychiatric hospital, 1st Psychogeriatric Department, Thessaloniki
  - Psychiatric Hospital of Thessaloniki, Psychiatric Department, Thessaloniki
  - G. Papanikolaou Hospital 3rd Neurology Clinic, Thessaloniki
  - Centre of Psychiatric Health, Tripoli

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2501054&StudyName=Quality%20Of%20Life%20Assesment%20In%20Alzheimer%27s%20Disease%20%28AD%29%20Patients%20Receiving%20Aricept%20Tablets%20

RESULTS

PARTICIPANT FLOW:
Groups:
- ARICEPT: ARICEPT (donepezil hydrochloride) 5 milligram (mg) or 10 mg once daily (QD) orally. 5 mg QD was maintained for at least 4 weeks. The recommended maximum dose was 10 mg QD.
Period: Overall Study
Arm/Group | ARICEPT
Started | 603
Completed | 573 (1 subject died during the study; 1 subject died following permanent discontinuation from the study.)
Not Completed | 30
Not completed — Death | 2
Not completed — Adverse Event | 15
Not completed — Lost to Follow-up | 8
Not completed — Other | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | ARICEPT
Number analyzed (Participants) | 603
Age, Customized [Number; unit: participants]
  18 to 44 years | 6
  45 to 64 years | 44
  65 years or older | 543
  Unspecified | 10
Sex/Gender, Customized [Number; unit: participants]
  Female | 364
  Male | 238
  Unspecified | 1
Medical History [Number; unit: participants] — Participants were counted once per medical history but could be counted in more than one medical history.
  participants
    Anaemia | 4
    Iron deficiency anaemia | 3
    Aortic valve incompetence | 1
    Arrhythmia | 1
    Atrial fibrillation | 7
    Cardiac failure | 1
    Coronary artery disease | 64
    Thalassaemia trait | 1
    Vertigo | 4
    Goitre | 3
    Hyperthyroidism | 7
    Hypothyroidism | 16
    Cataract | 4
    Eye disorder | 1
    Glaucoma | 1
    Colitis | 1
    Diverticulum | 1
    Diverticulum intestinal | 1
    Gastrooesophageal reflux disease | 3
    Pancreatitis chronic | 1
    Necrosis | 1
    Sarcoidosis | 1
    Erysipelas | 1
    Panencephalitis | 1
    Traumatic brain injury | 1
    Vitamin B12 decreased | 1
    Diabetes mellitus | 89
    Dyslipidaemia | 1
    Hypercholesterolaemia | 2
    Hyperlipidaemia | 129
    Hyperuricaemia | 3
    Arthritis | 2
    Arthropathy | 1
    Musculoskeletal pain | 1
    Osteoarthritis | 4
    Osteoporosis | 33
    Rheumatoid arthritis | 3
    Haemangioma | 1
    Prostate cancer | 3
    Carotid artery disease | 1
    Cerebral ischaemia | 51
    Cerebrovascular accident | 16
    Dementia | 2
    Diabetic neuropathy | 1
    Dystonia | 1
    Epilepsy | 7
    Extrapyramidal disorder | 3
    Headache | 1
    Migraine | 2
    Motor neurone disease | 1
    Multiple sclerosis | 2
    Myasthenia gravis | 1
    Parkinson's disease | 16
    Polyneuropathy | 2
    Sciatica | 2
    Tremor | 1
    Abnormal behaviour | 2
    Anxiety disorder | 3
    Bipolar disorder | 1
    Depression | 116
    Neurosis | 2
    Personality change due to a general medical condit | 1
    Phobia | 1
    Psychotic disorder | 3
    Psychotic disorder due to a general medical condit | 2
    Schizophrenia | 11
    Schizophrenia, paranoid type | 1
    Sleep disorder | 3
    Stress | 2
    Glomerulonephritis | 1
    Incontinence | 1
    Renal failure | 1
    Renal failure chronic | 2
    Urinary incontinence | 2
    Urinary retention | 1
    Benign prostatic hyperplasia | 9
    Prostatic disorder | 1
    Prostatomegaly | 9
    Asthma | 4
    Chronic obstructive pulmonary disease | 13
    Lichen sclerosus | 1
    Cardiac operation | 1
    Cardiac pacemaker insertion | 1
    Oesophageal operation | 1
    Arterial disorder | 1
    Hypertension | 273
    Temporal arteritis | 1
    Varicose vein | 1
    Venous insufficiency | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Change From Baseline for Clinical Global Impressions of Improvement (CGI-I) at Week 12
Description: CGI-I is a 7-point physician rated scale ranging from very much improved to very much worse.
Time Frame: Baseline, Week 12.
Population: Full Analysis Set (FAS): all enrolled participants who received at least 1 dose (including partial doses) of ARICEPT.
Measure: Number; unit: participants
Arm/Group | ARICEPT
Number analyzed (Participants) | 603
participants
  Missing | 26
  Not assessed | 5
  Very much improved | 27
  Much improved | 103
  Minimally improved | 277
  No change | 142
  Minimally worse | 20
  Much worse | 3
  Very much worse | 0
Statistical Analysis 1: Comparison: ARICEPT; The effect of possible prognostic factors response on response rate: primary diagnosis severity. Participants were classified as responders if they were very much improved or much improved from baseline; Test type: Superiority or Other; p = 0.0023, Regression, Logistic

2. Primary Outcome: Number of Participants for Change From Baseline for the Caregiver's Assessment of Improvement at Week 12
Description: The caregiver's assessment improvement was a 5-point rated scale ranging from much improved to much worse to the question 'compared to the severity of your relative's condition at baseline, how much do you feel it has changed?'.
Time Frame: Baseline, Week 12.
Population: FAS.
Measure: Number; unit: participants
Arm/Group | ARICEPT
Number analyzed (Participants) | 603
participants
  Missing | 39
  Much improved | 54
  Improved | 343
  No change | 140
  Worse | 27
  Much worse | 0
Statistical Analysis 1: Comparison: ARICEPT; The effect of possible prognostic factors on response: significant medical history. Participants were classified as responders if they were much improved or improved from baseline; Test type: Superiority or Other; p = 0.0382, Regression, Logistic

3. Primary Outcome: Change From Baseline in the Participant's Assessment for Quality of Life for Alzheimer's Dementia (QoL-AD) Overall and Subscale Scores at Week 12
Description: QoL-AD was comprised of 13 individual items, each measured on a 4-point Likert scale (ranging from 1 [poor] to 4 [excellent]). Overall QoL-AD score was the sum of the scores for the 13 individual items and ranged from 13 to 52, with higher scores indicating a higher health related quality of life.
Time Frame: Baseline, Week 12.
Population: FAS; (n)=number of participants evaluable at baseline and Week 12.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ARICEPT
Number analyzed (Participants) | 581
scores on a scale
  Physical health | 0.1 (0.51)
  Energy | 0.2 (0.58)
  Mood | 0.3 (0.70)
  Living situation | 0.2 (0.58)
  Memory | 0.3 (0.61)
  Family | 0.1 (0.56)
  Marriage | 0.1 (0.55)
  Friends | 0.1 (0.63)
  Self as a whole | 0.1 (0.57)
  Ability to do chores around the house | 0.2 (0.69)
  Ability to do things for fun | 0.3 (0.63)
  Money | 0.1 (0.57)
  Life as a whole | 0.2 (0.59)
  Overall score | 2.3 (4.33)
Statistical Analysis 1: Comparison: ARICEPT; The effect of possible prognostic factors on response: primary diagnosis severity; Test type: Superiority or Other; p = 0.1805, Regression, Linear
Statistical Analysis 2: Comparison: ARICEPT; The effect of possible prognostic factors on response: baseline QoL-AD score as assessed by participant; Test type: Superiority or Other; p < 0.0001, Regression, Linear
Statistical Analysis 3: Comparison: ARICEPT; The effect of possible prognostic factors on response: center number; Test type: Superiority or Other; p < 0.0001, Regression, Linear

4. Primary Outcome: Change From Baseline in the Caregiver's Assessment for Quality of Life for Alzheimer's Dementia (QoL-AD) Overall and Subscale Scores at Week 12
Description: as for outcome 3
Time Frame: Baseline, Week 12.
Population: FAS; (n)=number of participants evaluable at baseline and Week 12.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ARICEPT
Number analyzed (Participants) | 564
scores on a scale
  Physical health | 0.1 (0.54)
  Energy | 0.2 (0.65)
  Mood | 0.3 (0.72)
  Living situation | 0.2 (0.62)
  Memory | 0.3 (0.67)
  Family | 0.1 (0.52)
  Marriage | 0.1 (0.58)
  Friends | 0.1 (0.63)
  Self as a whole | 0.1 (0.63)
  Ability to do chores around the house | 0.2 (0.66)
  Ability to do things for fun | 0.2 (0.66)
  Money | 0.1 (0.62)
  Life as a whole | 0.1 (0.53)
  Overall score | 2.0 (4.58)
Statistical Analysis 1: Comparison: ARICEPT; The effect of possible prognostic factors on response: primary diagnosis severity; Test type: Superiority or Other; p = 0.0137, Regression, Linear
Statistical Analysis 2: Comparison: ARICEPT; The effect of possible prognostic factors on response: baseline QoL-AD score as assessed by caregiver; Test type: Superiority or Other; p < 0.0001, Regression, Linear
Statistical Analysis 3: Comparison: ARICEPT; The effect of possible prognostic factors on response: center number; Test type: Superiority or Other; p < 0.0001, Regression, Linear

5. Secondary Outcome: Change in ARICEPT Dosing: Number of Participants for Time to First ARICEPT Dose Escalation
Description: The starting dose of ARICPET was 5 mg once daily (QD), which could be increased to 10 mg QD during the study.
Time Frame: Baseline to Week 12.
Population: FAS. Starting dose of ARICEPT was not summarized.
Measure: Number; unit: participants
Arm/Group | ARICEPT
Number analyzed (Participants) | 603
participants
  Missing | 198
  0 weeks up to less than 4 weeks | 77
  4 weeks up to less than 6 weeks | 267
  6 weeks up to less than 8 weeks | 19
  8 weeks up to less than 10 weeks | 13
  10 weeks or later | 29

6. Secondary Outcome: Change in ARICEPT Dosing: Number of Participants at Each Final Dose of ARICEPT
Time Frame: Week 12.
Population: FAS.
Measure: Number; unit: participants
Arm/Group | ARICEPT
Number analyzed (Participants) | 603
participants
  Missing | 8
  5 mg | 193
  10 mg | 400
  greater than 10 mg | 2

7. Secondary Outcome: Number of Participants for the Physician's Assessment of Tolerance to ARICEPT at Week 12
Description: The physician rated tolerance to ARICEPT as very good, good, adequate, unsatisfactory, or unevaluable.
Time Frame: Baseline to Week 12.
Population: FAS.
Measure: Number; unit: participants
Arm/Group | ARICEPT
Number analyzed (Participants) | 603
participants
  Missing | 9
  Very good | 386
  Good | 161
  Adequate | 26
  Unstatisfactory | 13
  Unevaluable | 8

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | ARICEPT
Serious Adverse Events (participants affected / at risk) | 2/603
Other Adverse Events (participants affected / at risk) | 39/603
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARICEPT (N=603)
Death (General disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARICEPT (N=603)
Bradycardia (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
International normalised ratio increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 6
Psychomotor hyperactivity (Nervous system disorders) | 1
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 2
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Delusional disorder, unspecified type (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Dysthymic disorder (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Illusion (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.